CLINICAL TRIAL: NCT05047341
Title: A Clinical Trial of the Absorption, Metabolism and Excretion of [14C]SHR0302 in Healthy Chinese Adult Male Subjects
Brief Title: A Study of Human Substance Balance and Biotransformation of [14C]SHR0302
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR0302-107
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: This is a single-arm and open-label drug interaction study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: SHR0302、[14C]SHR0302

INTERVENTIONS:
Drug: SHR0302、[14C]SHR0302 — 8 mg SHR0302/ 80 µCi [14C]SHR0302, once, D1

SUMMARY:
The study is being conducted to evaluate the absorption, metabolism and excretion of [14C]SHR0302 in healthy Chinese adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, communicate well with the investigator and be able to complete the trial in strict compliance with the protocol;
2. Chinese male subjects judged by the investigator to be healthy;
3. Adults aged 18 to 45 years (including both ends of the spectrum, as at the time of signing the informed consent form);
4. Weight ≥ 50 kg and a body mass index (BMI) in the range of 19 to 26 kg/m2 (both ends inclusive).

Exclusion Criteria:

Ancillary examinations :

1. Abnormalities in physical examination, vital signs, routine laboratory tests (complete blood cell analysis, blood biochemistry, coagulation, urine routine, stool routine + occult blood), thyroid function, 12-lead ECG, chest CT, abdominal ultrasound (liver, gallbladder, pancreas, spleen and kidney) and other tests of clinical significance.
2. Resting corrected QT interval (QTcF) >450 ms obtained on a 12-lead ECG.
3. Positive for hepatitis B surface antigen or E antigen, hepatitis C antibody, HIV antibody and syphilis antibody.
4. Screening for novel coronavirus infection with clinically significant abnormal C-reactive protein or positive novel coronavirus nucleic acid.

   Medication history：
5. Systemic use of any drug that inhibits or induces CYP3A within 30 days prior to the screening period (e.g., inducers - bosentan, paracetamol, efavirenz, etravirine, phenobarbital, rifampin, mitotane, phenytoin sodium, carbamazepine, apatamide, etc.; inhibitors - -erythromycin, clarithromycin, fluconazole, ketoconazole, itraconazole, posaconazole, voriconazole, ciprofloxacin, diltiazem, fluvoxamine, nelfinavir, conivaptan, aripitant, crizotinib, imatinib, dronedarone, cyclosporine).
6. Have used any prescription drugs, over-the-counter medicines, herbal remedies or dietary supplements such as vitamins, calcium supplements within 14 days prior to the screening period.

   Medical and surgery history：
7. History of any clinically significant illness or disease or condition that, in the opinion of the investigator, may affect the results of the test, including but not limited to circulatory, respiratory, endocrine, neurological, digestive, urinary or haematological, immunological, psychiatric and metabolic disorders.
8. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmias, torsional ventricular tachycardia, ventricular tachycardia, atrioventricular block, QT prolongation syndrome or symptoms of QT prolongation syndrome and family history (indicated by genetic evidence or sudden death of a close relative at a young age due to cardiac causes).
9. Have undergone major surgery within the 6 months prior to the screening period or where the surgical incision has not fully healed; major surgery includes, but is not limited to, any surgery with significant risk of bleeding, extended general anaesthesia, or incisional biopsy or significant traumatic injury.
10. Allergies, such as a known history of allergy to two or more substances; or a potential allergy to the test drug or its excipients as judged by the investigator.
11. Haemorrhoids or perianal disease with regular/ongoing blood in the stool, irritable bowel syndrome, inflammatory bowel disease.

    Living habits：
12. Habitual constipation or diarrhoea.
13. Alcohol abuse or regular alcohol consumption within the 6 months prior to the screening period, i.e. more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits at 40% alcohol by volume or 150 mL of wine); or an alcohol breath test result of ≥20 mg/dL at the screening period.
14. Those who smoked more than 5 cigarettes per day or habitually used nicotine-containing products in the 3 months prior to the screening period and were unable to quit during the trial.
15. Substance abuse or use of soft drugs (e.g. cannabis) 3 months prior to the screening period or hard drugs (e.g. cocaine, amphetamines, phencyclidine, etc.) 1 year prior to the screening period; or a positive urine drug test during the screening period.
16. Habitual consumption of grapefruit juice or excessive amounts of tea, coffee and/or caffeinated beverages that cannot be abstained from during the trial.

    Others：
17. Workers exposed to prolonged radiological conditions; or who have had significant radiological exposure (≥2 chest/abdominal CTs, or ≥3 other types of X-ray examinations) or participated in radiopharmaceutical labelling tests within 1 year prior to the test.
18. People who have a history of needle sickness or blood sickness, have difficulty collecting blood or cannot tolerate venipuncture blood collection.
19. Participation in any other clinical trial (including clinical trials such as drugs and devices) within 3 months prior to the screening period.
20. Those who have been vaccinated within 1 month prior to screening or those who are scheduled to be vaccinated during the trial period.
21. Those who plan to have children or donate sperm during the trial and within 1 year after completion of the trial, or who do not agree that subjects and their spouses should use strict contraception during the trial and within 1 year after completion of the trial (see Annex 1 for details).
22. Those who have lost or donated up to 400 mL of blood within 3 months prior to the screening period, or those who have received a blood transfusion within 1 month.
23. Subjects who, in the opinion of the investigator, have any factors that make them unsuitable for this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Cmax | day 1 to day 11
AUC0-t | day 1 to day 11
AUC0-∞ | day 1 to day 11
Tmax | day 1 to day 11
t1/2 | day 1 to day 11
CL/F | day 1 to day 11
Vz/F | day 1 to day 11

SECONDARY OUTCOMES:
The incidence and severity of adverse events/serious adverse events | from ICF signing date to approximate day 11

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided